CLINICAL TRIAL: NCT01343251
Title: Prospective Analysis of Hemodialysis Reliable Outflow (HeRO) Vascular Access Graft vs. Cuffed Catheter Access in Hemodialysis
Brief Title: HeRO Graft Compared to Permanent Catheters for End Stage Renal Disease (ESRD) Patients Receiving Hemodialysis
Status: Completed | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HeRO-1
Record Dates: First submitted 2011-04-20; First posted 2011-04-28 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: dialysis; HeRO graft; catheter; chronic renal failure; end stage renal disease; renal insufficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HeRO Graft: patients who are evaluated and receive a HeRO Graft implant for hemodialysis
- Control: control group of non-HeRO patients who are evaluated but do not receive a HeRO Graft for any reason

SUMMARY:
The main objective of this research study was to compare the following outcomes between patients with a Hemodialysis Reliable Outflow (HeRO) Graft and patients with a cuffed catheter for dialysis access over one year: quality of life and incidence of bacteremia, vascular interventions, hospitalizations, and death.

DETAILED DESCRIPTION:
All eligible participants who provided informed consent were included in the study. Participants who refused HeRO Graft implantation, or did not have the HeRO Graft implanted for any other reason, were followed in the control group. Several patients did not receive the HeRO graft due to anatomical challenges and failure to complete both steps of the two-stage implant procedure. All consented participants who had an implanted HeRO Graft were followed in the study group. All participants were followed until the study end, withdrawal, loss to follow-up, or death. The analysis included only HeRO Graft patients and control patients who were not lost to follow-up; patients who were lost to follow-up, before data collection, were excluded from analysis.

After obtaining Institutional Review Board (IRB) approval, baseline demographic and clinical data was collected. Following surgery, implant procedure data was collected on study participants who received HeRO Grafts. HeRO Grafts were placed using a 2-step process with initial placement of the ePTFE portion, followed by completion of the graft by placement of the venous outflow component. Following enrollment, outcomes of interest were collected at follow-up visits scheduled weekly for 4 weeks, bi-weekly for 3 months, and monthly to 1 year, for a total of 18 follow-up visits. Study coordinators documented post-operative complications, incidence of thrombosis, hospitalizations, infection incidents, and deaths at each follow-up.

Quality of life data were also collected from all participants using the RAND Corporation's Short Form (36) (SF-36) Health Survey. This survey was completed at enrollment and again at 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients requiring hemodialysis
* Age ≥ 18 years old
* Able to give informed consent
* Able to participate in quality of life survey
* All patients who are not candidate for arteriovenous fistula (AVF) or arteriovenous graft (AVG)
* Life expectancy 2 years or greater
* Willing and able to participate with follow-up examinations

Exclusion Criteria:

* Pregnant or breastfeeding females
* Disorder that compromises the ability to give informed consent and/or comply with the study procedures
* Any medical condition that in the opinion of the investigator may pose a safety risk to a subject in the study or which may interfere with the study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ESRD requiring permanent cuffed catheters were targeted. Participants who had not exhausted peripheral venous access sites suitable for fistulas and grafts were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Provenzano, MD, Principal Investigator — St. Clair Specialty Physicians
Locations (1):
- St. Clair Specialty Physicians, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ethier J, Mendelssohn DC, Elder SJ, Hasegawa T, Akizawa T, Akiba T, Canaud BJ, Pisoni RL. Vascular access use and outcomes: an international perspective from the Dialysis Outcomes and Practice Patterns Study. Nephrol Dial Transplant. 2008 Oct;23(10):3219-26. doi: 10.1093/ndt/gfn261. Epub 2008 May 29. PMID 18511606
- [Background] Foley RN, Chen SC, Collins AJ. Hemodialysis access at initiation in the United States, 2005 to 2007: still "catheter first". Hemodial Int. 2009 Oct;13(4):533-42. doi: 10.1111/j.1542-4758.2009.00396.x. Epub 2009 Sep 16. PMID 19758304
- [Background] Mokrzycki MH, Zhang M, Cohen H, Golestaneh L, Laut JM, Rosenberg SO. Tunnelled haemodialysis catheter bacteraemia: risk factors for bacteraemia recurrence, infectious complications and mortality. Nephrol Dial Transplant. 2006 Apr;21(4):1024-31. doi: 10.1093/ndt/gfi104. Epub 2006 Jan 31. PMID 16449293
- [Background] Katzman HE, McLafferty RB, Ross JR, Glickman MH, Peden EK, Lawson JH. Initial experience and outcome of a new hemodialysis access device for catheter-dependent patients. J Vasc Surg. 2009 Sep;50(3):600-7, 607.e1. doi: 10.1016/j.jvs.2009.04.014. Epub 2009 Jul 22. PMID 19628360
- [Background] Hakim RM, Himmelfarb J. Hemodialysis access failure: a call to action--revisited. Kidney Int. 2009 Nov;76(10):1040-8. doi: 10.1038/ki.2009.318. Epub 2009 Aug 26. PMID 19710629
- [Background] Pisoni RL, Young EW, Dykstra DM, Greenwood RN, Hecking E, Gillespie B, Wolfe RA, Goodkin DA, Held PJ. Vascular access use in Europe and the United States: results from the DOPPS. Kidney Int. 2002 Jan;61(1):305-16. doi: 10.1046/j.1523-1755.2002.00117.x. PMID 11786113
- [Background] Surratt RS, Picus D, Hicks ME, Darcy MD, Kleinhoffer M, Jendrisak M. The importance of preoperative evaluation of the subclavian vein in dialysis access planning. AJR Am J Roentgenol. 1991 Mar;156(3):623-5. doi: 10.2214/ajr.156.3.1781814.
- [Background] Bohlke M, Uliano G, Barcellos FC. Hemodialysis catheter-related infection: prophylaxis, diagnosis and treatment. J Vasc Access. 2015 Sep-Oct;16(5):347-55. doi: 10.5301/jva.5000368. Epub 2015 Apr 20. PMID 25907773
- [Background] Yoon WJ, Lorelli DR. Avoiding the use of a femoral bridging catheter using a two-stage Hemodialysis Reliable Outflow (HeRO) graft implantation technique. J Vasc Access. 2015 May-Jun;16(3):189-94. doi: 10.5301/jva.5000325. Epub 2015 Jan 20. PMID 25613143
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Gage SM, Katzman HE, Ross JR, Hohmann SE, Sharpe CA, Butterly DW, Lawson JH. Multi-center experience of 164 consecutive Hemodialysis Reliable Outflow [HeRO] graft implants for hemodialysis treatment. Eur J Vasc Endovasc Surg. 2012 Jul;44(1):93-9. doi: 10.1016/j.ejvs.2012.04.011. Epub 2012 May 12. PMID 22580402
- [Background] Tonnessen BH, Money SR. Embracing the fistula first national vascular access improvement initiative. J Vasc Surg. 2005 Sep;42(3):585-6. doi: 10.1016/j.jvs.2005.05.030. No abstract available. PMID 16171614
- [Background] Berwick DM, Nolan TW, Whittington J. The triple aim: care, health, and cost. Health Aff (Millwood). 2008 May-Jun;27(3):759-69. doi: 10.1377/hlthaff.27.3.759. PMID 18474969
- [Background] Dageforde LA, Bream PR, Moore DE. Hemodialysis Reliable Outflow (HeRO) device in end-stage dialysis access: a decision analysis model. J Surg Res. 2012 Sep;177(1):165-71. doi: 10.1016/j.jss.2012.04.041. Epub 2012 May 9. PMID 22608835
- [Background] Ware JE, Kosinski M, Gandek. SF-36 Health Survey Manual & Interpretation Guide. Lincoln RI, Quality Metric Incorporated, 2000, pp. 10-14

RESULTS

PARTICIPANT FLOW:
Groups:
- HeRO Graft: patients who are evaluated and receive a Hemodialysis Reliable Outflow (HeRO) graft implant for hemodialysis
Period: Overall Study
Arm/Group | HeRO Graft | Control
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HeRO Graft | Control | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.69 (11.08) | 63.12 (11.49) | 60.00 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Compare mortality rate between study arms
Time Frame: 1 year
Measure: Number; unit: percentage of participants who died
Groups:
- HeRO Graft: HeRO Graft Recipients
- Control: HeRO eligible patients who did not receive HeRO
Arm/Group | HeRO Graft | Control
Number analyzed (Participants) | 16 | 17
percentage of participants who died | 18.8 | 29.4
Statistical Analysis 1: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p = 0.48, Chi-squared

2. Secondary Outcome: Infection Rate (Percentage of Participants With at Least One Infection)
Description: Compare incidence of infection between study arms
Time Frame: 1 year
Measure: Number; unit: Percentage of Patients
Arm/Group | HeRO Graft | Control
Number analyzed (Participants) | 16 | 17
Percentage of Patients | 25.0 | 64.7
Statistical Analysis 1: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p = 0.02, Chi-squared

3. Secondary Outcome: Quality of Life
Description: Compare the RAND Short Form (SF)-36 Health Survey, Total Test Scores at baseline, 3, 6, and 12 months between study arms. Total test scores range on a scale from 0-100, with the lower the score equating to more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. The total score is calculated using a methodology described by the RAND Corporation, which assigns a recoded value to each survey item. Recoded items are averaged amongst scales and the total score is an average of the eight sections. (http://www.rand.org/content/dam/rand/www/external/health/surveys_tools/mos/mos_core_36item_scoring.pdf).
Time Frame: 1 year
Population: The number of completed tests varied by time point and study group. The number of completed tests for Test 1, Test 2, Test 3, and Test 4 was 14, 13, 10, and 8 for the HeRO Graft group and 17, 13, 7, and 4 for the Control group, respectively. Only completed tests were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: HeRO eligible patients who did not receive a HeRO
Arm/Group | HeRO Graft | Control
Number analyzed (Participants) | 16 | 17
units on a scale
  Test 1 (Baseline) | 58.06 (25.49) | 51.30 (28.78)
  Test 2 (3 Months) | 56.30 (23.78) | 55.22 (22.40)
  Test 3 (6 Months) | 58.44 (22.08) | 53.53 (23.49)
  Test 4 (12 Months) | 60.41 (18.06) | 20.14 (4.67)
Statistical Analysis 1: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p = 0.49, t-test, 2 sided — SF-36 Test 1 Total Score
Statistical Analysis 2: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p = 0.91, t-test, 2 sided — SF-36 Test 2 Total Score
Statistical Analysis 3: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p = 0.67, t-test, 2 sided — SF-36 Test 3 Total Score
Statistical Analysis 4: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — SF-36 Test 4 Total Score

4. Secondary Outcome: Intervention Rate (Percentage of Participants Who Required at Least One Intervention While on Study)
Description: Compare vascular intervention rates between study arms. The vascular interventions which were included were: Angioplasty, Thrombectomy, Arteriovenous (AV) Fistulogram/Diagnostic Angiogram, Banding, Access Removal, Access Exchange, Access Revision, Creation of New Access, and any combination of these interventions which were performed simultaneously.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Groups:
- Control: HeRO eligible patients who did not receive a HeRO Graft
Arm/Group | HeRO Graft | Control
Number analyzed (Participants) | 16 | 17
percentage of participants | 93.8 | 64.7
Statistical Analysis 1: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p = 0.04, Chi-squared

5. Secondary Outcome: Hospitalization Rate (Percentage of Participants Who Were Hospitalized at Least Once While on Study)
Description: Compare incidence of hospitalization (for any reason) between study arms. Reasons for hospitalizations included: infection, cardiac problems, bleeding, vascular access thrombosis, fall (injury), hematuria, fluid overload, peripheral neuropathy, pulmonary embolism, edema, and shortness of breath.
Time Frame: 1 year
Measure: Number; unit: Percentage of patients
Arm/Group | HeRO Graft | Control
Number analyzed (Participants) | 16 | 17
Percentage of patients | 62.5 | 64.7
Statistical Analysis 1: Comparison: HeRO Graft vs Control; Test type: Superiority or Other; p = 0.90, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HeRO Graft | Control
Serious Adverse Events (participants affected / at risk) | 16/16 | 15/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeRO Graft (N=16) | Control (N=17)
Bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arteriosclerotic Heart Disease (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (3)
Pulmonary Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death-Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Death-Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Death-Unknown Cause (General disorders) | 3 (3) | 3 (3)
Infection (Infections and infestations) | 6 (11) | 12 (18)
Injury-Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Fluid Overload (Renal and urinary disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Access Creation (Vascular disorders) | 0 (0) | 3 (3)
Access Exchange (Vascular disorders) | 1 (2) | 4 (9)
Access Explant (Vascular disorders) | 2 (3) | 0 (0)
Access Revision (Vascular disorders) | 1 (1) | 1 (1)
Graft Swelling (Vascular disorders) | 1 (1) | 0 (0)
Intervention to Restore Patency (Vascular disorders) | 12 (35) | 4 (5)
Pseudoaneurysm (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Target sample size (statistical power) was not achieved. Catheter reduction and fistula first policies limited recruitment. Additionally, study patients were not blind to exposure and this knowledge may have had an impact on QoL measurement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No